CLINICAL TRIAL: NCT00015600
Title: Community-Based Environmental Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8766-CP-001
Record Dates: First submitted 2001-04-23; First posted 2001-04-25 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Poisoning
Keywords: Pesticide; Farmworker; Occupational health
MeSH Terms: conditions — Poisoning

INTERVENTIONS:
Behavioral: Behavior modification through social marketing

SUMMARY:
This community-based project, called the Together for Agricultural Safety project, was developed to help farmworkers reduce their exposure to dangerous agricultural chemicals (such as pesticides) through education and social marketing. The project is a partnership of university researchers and the Farmworkers Association of Florida. After collecting extensive data from farmworkers, health providers and farm owners about primary means of pesticide exposure we are collaboratively developing an intervention that will reduce pesticide exposure by educating workers and owners about: the need to have adequate washing facilities; to wash hands frequently; to obey reentry intervals; to change work clothes after work to prevent child exposure and more.

ELIGIBILITY:
Must be an agricultural worker in the fernery or nursery industries in Central Florida.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1997-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States